CLINICAL TRIAL: NCT01022138
Title: A Phase II Study of Anti-CD3 x Anti-HER2/Neu Armed Activated T Cells for Patients With HER2/Neu (0, 1+ or 2+) Metastatic Breast Cancers.
Brief Title: Laboratory-Treated T Cells After Second-Line Chemotherapy in Treating Patients With HER2/Neu-Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abhinav Deol, Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-085; P30CA022453 (NIH); WSU-2009-085 (Other: Karmanos Cancer Center)
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: HER2-negative breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HER2Bi-armed activated T cells/Cyclophosphamide/biomarker (Experimental): HER2Bi-armed activated T cells Immediately after pheresis, the lymphocytes are activated with soluble monoclonal anti-CD3 antibody, which cross-links the CD3 receptors on T cells and activates them.
  Cyclophosphamide After recovering from the last cycle of chemotherapy (approx. two-four weeks) patients will be re-staged. If there are no residual chemotherapy related toxicities, they will be given lymphodepleting chemotherapy consisting of one dose of Cyclophosphamide 1.0 gm/m2 on day -7. Appropriate anti-emetics will be given as pre-medications before the dose of Cyclophosphamide
  Laboratory biomarker analysis The association between the [18F]-FDG PET/CT assessments (percent changes from baseline in SUVpeak) and immunologic biomarker changes as well as tumor response will be explored.
  Interventions: Biological: HER2Bi-armed activated T cells; Drug: Cyclophosphamide; Other: Laboratory biomarker analysis

INTERVENTIONS:
Biological: HER2Bi-armed activated T cells — Immediately after pheresis, the lymphocytes are activated with soluble monoclonal anti-CD3 antibody, which cross-links the CD3 receptors on T cells and activates them.
Drug: Cyclophosphamide — After recovering from the last cycle of chemotherapy (approx. two-four weeks) patients will be re-staged. If there are no residual chemotherapy related toxicities, they will be given lymphodepleting chemotherapy consisting of one dose of Cyclophosphamide 1.0 gm/m2 on day -7. Appropriate anti-emetics will be given as pre-medications before the dose of Cyclophosphamide
Other: Laboratory biomarker analysis — The association between the [18F]-FDG PET/CT assessments (percent changes from baseline in SUVpeak) and immunologic biomarker changes as well as tumor response will be explored.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Treating a patient's T cells in the laboratory may help the T cells kill more tumor cells when they are put back in the body. Giving laboratory-treated T cells after chemotherapy may be an effective treatment for breast cancer.

PURPOSE: This phase II trial is studying how well giving laboratory-treated T cells after second-line chemotherapy works in treating patients with HER2/neu-negative metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine in a phase II trial whether Her2Bi armed ATC infused after ChemoT for patients with HER2 0-2+ MBC or locally advanced, unresectable breast cancer would improve median PFS by 2 months beyond the median PFS of 2 months estimated from published trials in a one stage design.
* To determine the overall survival (OS) of patients with HER2 0-2+ MBC and locally advanced, unresectable breast cancer who receive aATC infusion after ChemoT.
* To confirm the toxicity profile for Her2Bi armed ATC given after ChemoT for patients with HER2 0-2+ MBC.
* To measure functional and phenotypic changes in immune cell populations (blood and tumor sites, if accessible) as a consequence of armed ATC (tumor biopsies done at KCI only). Cytokine responses, phenotypic markers of differentiation, and anti-tumor cytotoxicity will be examined.
* OUTLINE: Patients receive second-line chemotherapy for 4 courses or 4 months. Beginning as early as 1.5 weeks and as late as 4 weeks after chemotherapy, the patients will receive the first infusion of anti-CD3 x anti-HER2/neu bispecific antibody-armed activated T-cells (ATC) IV over 30-60 minutes once a week for 3 weeks. Low dose granulocyte-macrophage colony stimulating factor (250 µg/m2/twice per week) will start 3 days before the first aATC infusion and end with the last dose of aATC. Patients who are already on the protocol will be given a choice to add GM-CSF to their treatment regimen (after reconsenting) or continue to their treatment without GM-CSF. Patients then receive a boost of anti-CD3 x anti-HER2/neu bispecific antibody-armed ATC at 12 weeks after the 3rd ATC infusion.

Blood and tumor tissue samples may be collected periodically for biomarker and other analyses.

After completion of study therapy, patients are followed up periodically for ≥ 2 years.

ELIGIBILITY:
Inclusion:

* Metastatic Breast Cancer. Histologically confirmed breast cancer with evidence of metastatic disease (need not be biopsy proven) or locally, advanced unresectable disease.
* Patients with 0-2+ HER2 expression as determined by immunohistochemistry staining and/or FISH ratio <2.0, with the above pathologic criteria will be eligible.
* Hormone Therapy. Patients on prior hormonal therapy are eligible. Hormonal therapy will be stopped 2 weeks prior to leukopheresis. Hormone therapy may be restarted after leukopheresis
* Patients may have received any number of prior lines of chemotherapy providing Leukopheresis is done when the lymphocyte count has recovered to ≥500 cells/mm3 and there are no residual chemotoxicities that would prevent leukopheresis.
* Patients who have received Radiotherapy are eligible providing Leukopheresis is done at least 4 weeks after radiation to the axial skeleton.
* Patients who have received prior biological agents are eligible.
* Patients with measurable and non-measurable disease are eligible.
* Age > or = to 18 years
* ECOG 0-1 or Karnofsky > or = to 70%
* Life expectancy > or = to 3 months
* Patients with treated brain metastases are eligible
* Required Laboratory Data Granulocytes > 1,200/mm3 Platelet count > 50,000/μl Hemoglobin ≥ 8 gm/dl BUN < 1.5 times normal Serum creatinine < 1.8 mg/dl Creatinine Cl ≥50 ml/mm (can be calculated utilizing the Cockcroft & Gault equation: Creatinine Clearance (mL/min) = {(140 - Age)} x Wt [kg] (x 0.85 if Female}/ {72 x SCr [mg/dL]} Bilirubin < 1.5 times normal ALT, AST and alkaline phosphatase < 5 times upper normal Negative HIV Negaitve Hepatitis B surface antigen Negative Hepatitis C serology LVEF ≥ 45% at rest (MUGA or ECHO) PFT-FEV1, DLCO, and FVC ≥ 50% of predicted
* Negative serum test for pregnancy, unless male, prior hysterectomy, tubal ligation, or postmenopausal. (Note: postmenopausal is defined as age>55 with amenorrhea for >1 year or age <55 years with amenorrhea for 2 years and FSH level within postmenopausal range of institutional parameters; patients requiring FSH level to determine menopausal status need not have this performed and may choose to proceed with serum pregnancy testing.)

Exclusion Criteria

* Patients with HER2 overexpression by immunohistochemistry (IHC) or overamplification by FISH are not eligible and are defined as follows: IHC staining of 3+ (uniform, intense membrane staining of > 30% of invasive tumor cells), a fluorescent in situ hybridization (FISH) result of more than six HER2 gene copies per nucleus or a FISH ratio (HER2 gene signals to chromosome 17 signals) of more than 2.0.
* Patients with a history of another malignancy within 5 years of study entry are not eligible (except basal cell skin carcinoma and carcinoma-in-situ of the cervix).
* No serious medical or psychiatric illness which prevents informed consent or intensive treatment is allowed.
* Patients will be ineligible for treatment on this protocol if (prior to protocol entry):

  * There is a history of a recent myocardial infarction (within one year)
  * There is a history of a past myocardial infarction (more than one year ago) along with current coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by MUGA or ECHO)
  * There is a current history of angina/coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by MUGA or ECHO)
  * There is clinical evidence of congestive heart failure requiring medical management (irrespective of MUGA or ECHO results)
* Patients will be ineligible if there is recurrent pleural effusion or ascites requiring drainage (through thoracentesis, paracentesis, or indwelling device) more often than once every 4 weeks.
* Patients with clinical evidence of active CNS metastases are ineligible for therapy on this protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-03-08 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Deol, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 2010-2014; Location: Karmanos Cancer Institute, Detroit, MI
Period: Overall Study
Arm/Group | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker
Started | 43
Completed | 31
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 53.0 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Who Were Alive Without Progression at 4 Months
Description: 26 evaluable patients will be accrued in this study. A single-arm, single-stage phase II design will be used. If ≥9 out of 26 patients have not progressed by the 4-month follow-up, we will declare that the treatment is effective on TTP.
Time Frame: At the 4-month follow-up
Population: There were 32 evaluable HER2 negative patients who received therapy out 42 female patients who were originally enrolled, where one male participant was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker: * HER2Bi-armed activated T cells: Immediately after pheresis, lymphocytes are activated with soluble monoclonal anti-CD3 antibody, which cross-links the CD3 receptors on T cells and activates them.
  * Cyclophosphamide: After recovering from last cycle of chemotherapy (approx. two-four weeks) patients will be restaged. If there is no residual chemotherapy related toxicities, they will be given lymphodepleting chemotherapy consisting of one dose of Cyclophosphamide 1.0 gm/m2 on day -7. Appropriate anti-emetics will be given as pre-medications before the dose of Cyclophosphamide
  * Laboratory biomarker analysis: Association between the [18F]-FDG PET/CT assessments (percent changes from baseline in SUVpeak) and immunologic biomarker changes as well as tumor response will be explored.
Arm/Group | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker
Number analyzed (Participants) | 32
Participants | 9

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time duration from the first infusion until death or last observation.
Time Frame: Followed until death or last observation (assessed up to 5 years), whichever occurs first
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker
Number analyzed (Participants) | 32
Months | 13.1 [8.6 to 17.4]

3. Secondary Outcome: Overall Response Rate
Description: Complete and partial responses; Responses will be evaluated using standard RECIST 1.1 criteria.
Time Frame: Following chemotherapy, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker
Number analyzed (Participants) | 32
Participants | 9

ADVERSE EVENTS:
Groups:
- HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker: HER2Bi-armed activated T cells Immediately after pheresis, the lymphocytes are activated with soluble monoclonal anti-CD3 antibody, which cross-links the CD3 receptors on T cells and activates them.
  Cyclophosphamide After recovering from the last cycle of chemotherapy (approx. two-four weeks) patients will be re-staged. If there are no residual chemotherapy related toxicities, they will be given lymphodepleting chemotherapy consisting of one dose of Cyclophosphamide 1.0 gm/m2 on day -7. Appropriate anti-emetics will be given as pre-medications before the dose of Cyclophosphamide
  Laboratory biomarker analysis The association between the [18F]-FDG PET/CT assessments (percent changes from baseline in SUVpeak) and immunologic biomarker changes as well as tumor response will be explored.
  HER2Bi-armed activated T cells: Immediately after pheresis, the lymphocytes are activated with soluble monoclonal anti-CD3 antibody, which cross-links the CD3 receptors on T cells and acti
Arm/Group | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker
All-Cause Mortality (participants affected / at risk) | 27/42
Serious Adverse Events (participants affected / at risk) | 6/42
Other Adverse Events (participants affected / at risk) | 32/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker (N=42)
Ascites (General disorders) | 1 (1)
AST, SGOT (General disorders) | 1 (1)
Leukocytes (General disorders) | 1 (1)
Cardiac General (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Somnolence/depressed level of consciousness (General disorders) | 1 (1)
Hypoxia (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Musculoskeletal/Soft Tissue (General disorders) | 1 (1)
Creatinine (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2Bi-armed Activated T Cells/Cyclophosphamide/Biomarker (N=42)
Ascites (General disorders) | 1 (3)
Chills (General disorders) | 30 (82)
Creatinine (General disorders) | 1 (1)
Diarrhea (General disorders) | 2 (2)
Dyspnea (General disorders) | 4 (5)
Fatigue (General disorders) | 31 (92)
Fever (General disorders) | 19 (38)
Headache (General disorders) | 22 (45)
Hypertension (General disorders) | 3 (4)
Hypoglycemia (General disorders) | 1 (1)
Hypotension (General disorders) | 14 (23)
Hypoxia (General disorders) | 2 (2)
Metabolic/Laboratory (General disorders) | 1 (2)
Muscle weakness (General disorders) | 1 (1)
Nausea (General disorders) | 20 (40)
Pain (General disorders) | 4 (5)
Somnolence (General disorders) | 1 (2)
Tachycardia (General disorders) | 2 (2)
Vomiting (General disorders) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT01022138/Prot_SAP_000.pdf